CLINICAL TRIAL: NCT02205814
Title: A Double-blind, Randomised, Placebo-controlled, Four Parallel Arm, Dose-finding Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Single Intra-articular Injections of Fasitibant in Patients With Symptomatic Osteoarthritis of the Knee.
Brief Title: Fasitibant Intra-articular Injection in Patients With Symptomatic Osteoarthritis of the Knee
Acronym: ALBATROSS-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BKOS-04; 2013-004999-35 (EudraCT Number)
Record Dates: First submitted 2014-07-14; First posted 2014-07-31 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis, Knee; Arthritis; WOMAC; Injections, intra-articular; Fasitibant; MEN 16132
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis | interventions — (4-amino-5-(4-(4-(2,4-dichloro-3-(2,4-dimethyl-8-quinolyloxymethyl)phenylsulfonamido)tetrahydro-2H-4-pyranoylcarbonyl)piperazino)-5-oxopentyl)(trimethyl)ammonium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fasitibant low dose (Experimental): Drug: solution for intra-articular injection
  Interventions: Drug: Fasitibant- low dose
- Fasitibant intermediate dose (Experimental): Drug: solution for intra-articular injection
  Interventions: Drug: Fasitibant- intermediate dose
- Fasitibant high dose (Experimental): Drug: solution for intra-articular injection
  Interventions: Drug: Fasitibant- high dose
- PLACEBO (Placebo Comparator): Drug: solution for intra-articular injection
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Fasitibant- low dose — Single intra-articular injection of low dose of fasitibant
  Arms: Fasitibant low dose
Drug: Fasitibant- intermediate dose — Single intra-articular injection of intermediate dose of fasitibant
  Arms: Fasitibant intermediate dose
Drug: Fasitibant- high dose — Single intra-articular injection of high dose of fasitibant
  Arms: Fasitibant high dose
Drug: Placebo comparator — Single intra-articular injection of placebo
  Arms: PLACEBO

SUMMARY:
This study is designed as a double-blind, randomised, placebo-controlled, four parallel arm, dose-finding study, to be conducted in approximately 26 sites, to evaluate the efficacy, safety, tolerability, and pharmacokinetics of single intra-articular (IA) injections of fasitibant in patients with symptomatic osteoarthritis (OA) of the knee.

Approximately 400 male and female patients 40-80 years old, with BMI < 30 kg/m² and with a clinical diagnosis of symptomatic primary osteoarthritis of the knee will be randomised to a total of 4 treatment arms. Each arm includes a single intra-articular injection of one of three dosages of fasitibant (low, intermediate and high dose) OR placebo. The randomisation ratio will be 1:1:1:1.

The primary efficacy variable will be the change of the Western Ontario and McMaster Universities Visual Analogue Scale 3.1 A (WOMAC VA 3.1 A) (total pain) subscore from baseline up to 2 weeks after randomisation. Safety will be assessed by monitoring adverse events and clinical laboratory tests; local tolerability at the injection site will also be assessed. In addition, the population pharmacokinetics and the exposure-response relationship will be evaluated.

The individual experimental clinical phase will last up to maximal 15 weeks encompassing 7 planned visits at site, including screening, randomisation, 4 follow-up visits and the End of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 40 to 80 years with BMI < 30 kg/m²
* Patient with Kellgren-Lawrence Grade 2 to 3, symptomatic primary osteoarthritis at the index knee (ACR criteria), for which an IA treatment is indicated
* Pain of moderate to severe intensity, even if treated with chronic doses of non steroidal antinflammatory drugs

Exclusion Criteria:

* History of hypersensitivity/allergy to drugs including paracetamol and to disinfectants
* Any pharmacological treatment of concomitant disease(s) started or changed during 4 weeks prior to randomisation, or likely to be changed during the course of the study
* Use of systemic or topical corticosteroids > 10 mg prednisolone equivalent per day, or immunosuppressant drugs
* Current use of any pain or OA medication (e.g. NSAIDs, COX-2 inhibitors, analgesics, antidepressive agents), including topical treatments
* Viscosupplementation to the target knee administered < 4 months prior to randomisation and/or scheduled during the course of the study
* Evidence of clinically significant hepatic disease or of moderate or severe renal insufficiency
* Current use of any medications that are substrate of CYP3A4 and/or moderate or strong CYP3A4 inhibitors
* Patients with any clinically relevant or unstable disease, or malignant neoplasms that, in the opinion of the Investigator, may pose the patient at risk, or confound the efficacy and safety results of the study
* Patients with any clinically relevant abnormal safety laboratory test results, and/or abnormalities in vital signs, and/or ECG parameters
* Pregnant and breastfeeding women
* Any sign of significant immunodeficiency, systemic infection, knee infection or knee bursitis
* Patients with bleeding diathesis or on therapy with anticoagulants

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karel Pavelka, Professor, Study Chair — Institute of Rheumatology, Charles University Faculty Hospital, Na Slupi 4, 128 50 Prague 2, Czech Republic
Locations (25):
- United States (9):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Colorado Orthopaedic Consultants, Englewood, Colorado
  - Avail Clinical Research, LLC, DeLand, Florida
  - Radiant Research, Columbus, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - Blair Orthopaedic Associates, Altoona, Pennsylvania
  - Tekton Research, Austin, Texas
  - Physicians Research Options, LLC, Draper, Utah
  - Spokan Joint Replacement Center, Spokane, Washington
- Czechia (3):
  - Revmatologie s.r.o., Brno
  - Institute of Rheumatology, Charles University Faculty Hospital, Prague
  - MEDICAL PLUS s.r.o, Uherské Hradiště
- Germany (6):
  - Synexus Clinical Research GmbH, Research Centre Berlin, Berlin
  - Synexus Clinical Research GmbH, Research Centre Bochum, Bochum
  - Synexus Clinical Research GmbH, Research Centre Frankfurt, Frankfurt
  - Clinical Research Hamburg GmbH, Hamburg
  - Synexus Clinical Research GmbH, Research Centre Leipzig, Leipzig
  - AmBeNet GmbH, Leipzig
- Italy (7):
  - Dipartimento di Medicina Interna - SOD di Reumatologia Azienda - Ospedaliero Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero-Universitaria S.Anna/ Unità Operativa Complessa e Sezione di Reumatologia/Dipartimento di Medicina Clinica e Sperimentale, Cona
  - Ospedale Galateo U.O. di Reumatologia, Lecce
  - Ospedale Fornaroli/Unità Complessa di Reumatologia, Magenta
  - Ospedale Luigi Sacco, Azienda Ospedaliera, Polo Universitario/Unità Operativa Complessa di Reumatologia, Milan
  - Azienda Ospedaliera di Perugia/Policlinico di Monteluce/Unità Operativa diagnosi e cura delle malattie reumatiche, Perugia
  - Centro Ricerche Cliniche di Verona, Verona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was screened on 28th April 2014. The first patient was randomised on 6th May 2014. The last patient completed the study on 6th January 2015.
  The study was conducted in 25 study sites in Czech Republic, Germany, Italy and US.
Pre-assignment Details: A total of 645 patients entered a 2-week Screening period (including wash out); 209 of them were screen failed. One patient randomised to PLACEBO did not receive the study treatment (counted for ITT but not in safety population). Five patients received the study treatment without randomisation (not counted for ITT, but in safety population).
Period: Overall Study
Arm/Group | Fasitibant Low Dose | Fasitibant Intermediate Dose | Fasitibant High Dose | PLACEBO
Started | 110 | 110 | 108 | 108
Completed | 108 | 109 | 103 | 104
Not Completed | 2 | 1 | 5 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1
Not completed — not compliant with study procedures | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on the ITT-population (n=431). The ITT-population included all patients randomised via IXRS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasitibant Low Dose | Fasitibant Intermediate Dose | Fasitibant High Dose | PLACEBO | Total
Number analyzed (Participants) | 108 | 108 | 107 | 108 | 431
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 65.3 (7.61) | 63.2 (8.73) | 64.7 (8.43) | 64.4 (8.50) | 64.4 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 71 | 64 | 66 | 263
  Male | 46 | 37 | 43 | 42 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 4
  Not Hispanic or Latino | 107 | 108 | 106 | 106 | 427
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.1 (2.12) | 26.5 (2.83) | 27.1 (2.35) | 27.0 (2.60) | 26.9 (2.50)
WOMAC A [Mean (Standard Deviation); unit: units on a scale] — The validated Western Ontario and McMaster University questionnaire (WOMAC) was used to measure total knee pain choosing its visual analogue scale version (VAS). The WOMAC VA 3.1 A subscore (WOMAC A) ranges from 0 to 500 mm (summing up five VAS 0-100 mm) with higher scores indicating more pain.
  units on a scale | 286.5 (40.4) | 282.7 (40.08) | 278.3 (38.11) | 275.5 (39.81) | 280.8 (39.61)
WOMAC INDEX [Mean (Standard Deviation); unit: units on a scale] — The WOMAC VA 3.1 Index score (WOMAC INDEX) is the sum of WOMAC A (total pain), WOMAC B (stiffness) and WOMAC C (functional impairment) subscores. The WOMAC INDEX score ranges from 0 to 2400 mm, with higher scores indicating higher disease burden.
  units on a scale | 1321.5 (278.88) | 1275.4 (283.60) | 1282.6 (274.50) | 1293.5 (239.73) | 1293.3 (269.35)
EQ VAS [Mean (Standard Deviation); unit: units on a scale] — The EQ visual analogue scale (EQ VAS) recorded the respondent's self-rated health on a 20 cm vertical VAS with endpoints labelled 'the best health you can imagine' on top (equal to 100) and 'the worst health you can imagine' at the bottom (equal to 0).
  units on a scale | 63.1 (20.54) | 64.3 (17.21) | 67.4 (18.18) | 65.7 (19.47) | 65.1 (18.89)

OUTCOME MEASURES:

1. Primary Outcome: Change in WOMAC A
Description: The validated Western Ontario and McMaster University questionnaire (WOMAC) was used to measure total knee pain choosing its visual analogue scale version (VAS). The WOMAC VA 3.1 A subscore (WOMAC A) ranges from 0 to 500 mm (summing up five VAS 0-100 mm) with higher scores indicating more pain.
Time Frame: from baseline up to 2 weeks after randomisation
Population: The primary efficacy analysis was performed on the ITT-population (n=431).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fasitibant Low Dose | Fasitibant Intermediate Dose | Fasitibant High Dose | PLACEBO
Number analyzed (Participants) | 108 | 108 | 107 | 108
units on a scale
  Week 1 after randomisation | -91.8 (101.85) | -110.0 (99.48) | -109.8 (94.65) | -93.7 (94.15)
  Week 2 after randomisation | -106.1 (101.88) | -131.5 (96.41) | -115.9 (104.61) | -117.2 (90.15)
Statistical Analysis 1: Comparison: Fasitibant Low Dose vs Fasitibant Intermediate Dose vs Fasitibant High Dose vs PLACEBO; Test type: Superiority or Other; p < 0.05, mixed linear model for repeated measures — Fourhundred evaluable patients were supposed to provide approximately 80% power in rejecting the null hypothesis of equality between any dose of fasitibant and placebo based on previous results and an overall significance level of 5% (two-sided)

2. Secondary Outcome: Change in WOMAC INDEX
Description: The WOMAC VA 3.1 Index score (WOMAC INDEX) is the sum of WOMAC A (total pain), WOMAC B (stiffness) and WOMAC C (functional impairment) subscores. The WOMAC INDEX score ranges from 0 to 2400 mm, with higher scores indicating higher disease burden.
Time Frame: from baseline up to 6 weeks after randomisation
Population: The secondary efficacy analysis was performed on the ITT population (n=431).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fasitibant Low Dose | Fasitibant Intermediate Dose | Fasitibant High Dose | PLACEBO
Number analyzed (Participants) | 108 | 108 | 107 | 108
units on a scale
  Week 1 after randomisation | -396.0 (464.24) | -460.5 (469.68) | -445.2 (424.07) | -413.2 (452.04)
  Week 2 after randomisation | -448.0 (477.95) | -563.0 (456.71) | -488.7 (480.39) | -517.7 (440.75)
  week 4 after randomisation | -516.4 (513.70) | -628.4 (500.17) | -493.4 (513.94) | -562.3 (487.25)
  Week 6 after randomisation | -566.3 (525.63) | -653.8 (516.31) | -547.6 (522.37) | -581.3 (503.37)
Statistical Analysis 1: Comparison: Fasitibant Low Dose vs Fasitibant Intermediate Dose vs Fasitibant High Dose vs PLACEBO; All secondary efficacy variables were analysed on the ITT population only. Multiplicity was adjusted using the Hochberg procedure. The continuous secondary efficacy variables were analysed over time and were treated in the same way as the primary efficacy variable with respective output; Test type: Superiority or Other; p < 0.05, mixed linear model for repeated measures — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Responder Rate According to OMERACT-OARSI Criteria
Description: Percentage of responders according to Outcome Measures in Rheumatology-Osteoarthritis Research Society International criteria (OMERACT-OARSI criteria). Patients with at least 50 % improvement in pain or in function scores are considered responders. Alternatively, patients are considered responders if they show at least 20% improvement in at least two of the following scores: pain, function and Patients's Global Assessment (PGA) scores.
Time Frame: from baseline up to 6 weeks after randomisation
Population: The secondary efficacy variables were analysed in the ITT population (n=431).
Measure: Number; unit: percentage of responders
Arm/Group | Fasitibant Low Dose | Fasitibant Intermediate Dose | Fasitibant High Dose | PLACEBO
Number analyzed (Participants) | 108 | 108 | 107 | 108
percentage of responders
  Week 1 after randomisation | 51.9 | 56.5 | 63.6 | 55.6
  Week 2 after randomisation | 59.3 | 72.2 | 62.6 | 68.5
  Week 4 after randomisation | 65.7 | 72.2 | 65.4 | 66.7
  Week 6 after randomisation | 71.3 | 74.1 | 67.3 | 67.6

4. Secondary Outcome: Euro Quality of Life Questionnaire (EQ-5D-5L) Responder Rate
Description: Response based on change ≥ 20 % from baseline for EQ-5D-5L index value
Time Frame: from baseline up to 6 weeks after randomisation
Population: The secondary efficacy analysis was performed on the ITT-population (n=431).
Measure: Number; unit: percentage of responders
Arm/Group | Fasitibant Low Dose | Fasitibant Intermediate Dose | Fasitibant High Dose | PLACEBO
Number analyzed (Participants) | 108 | 108 | 107 | 108
percentage of responders
  Week 2 after randomisation | 18.5 | 18.5 | 20.6 | 24.1
  Week 6 after randomisation | 23.1 | 27.8 | 25.2 | 21.3

ADVERSE EVENTS:
Time Frame: For all patients receiving the study treatment (safety population, N=435), adverse event data were collected over a period of maximal 15 weeks.
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Arm/Group | Fasitibant Low Dose | Fasitibant Intermediate Dose | Fasitibant High Dose | PLACEBO
Serious Adverse Events (participants affected / at risk) | 2/110 | 2/110 | 2/108 | 4/107
Other Adverse Events (participants affected / at risk) | 28/110 | 46/110 | 36/108 | 44/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasitibant Low Dose (N=110) | Fasitibant Intermediate Dose (N=110) | Fasitibant High Dose (N=108) | PLACEBO (N=107)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant breast lump removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasitibant Low Dose (N=110) | Fasitibant Intermediate Dose (N=110) | Fasitibant High Dose (N=108) | PLACEBO (N=107)
Nasopharyngitis (Infections and infestations) | 4 (4) | 17 (18) | 11 (11) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 7 (7) | 5 (6) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 5 (5) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 2 (3)
Injection site haematoma (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 3 (4) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the Investigator will allow the sponsor at least 30 days time to review and comment upon the publication manuscript. It is agreed, that the results of the study will not be submitted for presentation, abstract, poster exhibition, or publication by the investigator until the sponsor has reviewed/commented and agreed to any publication.